CLINICAL TRIAL: NCT01541995
Title: Evaluation of Contrast Medium Enhanced Post-mortem CT in Virtual Autopsy
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: VA-3 Contrast Medium
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Thromboembolism; Vascular Conditions
Keywords: contrast medium enhanced post mortem CT; virtual autopsy; To evaluate the value of contrast medium enhanced post-mortem CT in virtual autopsy focussing on thromboembolic and vascular conditions
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- virtual and classic autopsy: Patients where contrast medium enhanced post mortem CT and classic autopsy will be performed.
- virtual autopsy only: Patients where only contrast medium enhanced post mortem CT will be performed.

SUMMARY:
The study aims to compare the value of contrast medium enhanced post mortem CT to classic autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients dying in the ICU
* age >18y

Exclusion Criteria:

* relatives refusing to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients dying in the ICU during the study period
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Wichmann D, Heinemann A, Weinberg C, Vogel H, Hoepker WW, Grabherr S, Pueschel K, Kluge S. Virtual autopsy with multiphase postmortem computed tomographic angiography versus traditional medical autopsy to investigate unexpected deaths of hospitalized patients: a cohort study. Ann Intern Med. 2014 Apr 15;160(8):534-41. doi: 10.7326/M13-2211. PMID 24733194